CLINICAL TRIAL: NCT03279640
Title: Investigation for Individualized Noninvasive Neuromodulation in Neurorehabilitation of Brain Disease: Longitudinal Study
Brief Title: Effects of Brain Network by Simultaneous Dual-mode Stimulation in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-06-002
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-06

CONDITIONS: Stroke; Motor Disorder
Keywords: Motor Network; Resting-state fMRI; Repetitive Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Stroke; Motor Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-mode stimulation (Experimental): rTMS on ipsilesional M1 + tDCS on contralesional M1
  10 Hz of rTMS was applied over the ipsilesional M1 for 20 minutes with simultaneous application of cathodal tDCS on the contralesional M1.
  Each participant's total FMA score is assessed and their resting-state fMRI data at two times: prior to stimulation (pre-stimulation) and 2 months after stimulation (post-stimulation) are acquired.
  Interventions: Device: rTMS on ipsilesional M1; Device: tDCS on contralesional M1
- Single stimulation (Experimental): rTMS on ipsilesional M1
  10 Hz of rTMS over the ipsilesional M1 was applied for 20 minutes.
  Each participant's total FMA score is assessed and their resting-state fMRI data at two times: prior to stimulation (pre-stimulation) and 2 months after stimulation (post-stimulation) are acquired.
  Interventions: Device: rTMS on ipsilesional M1

INTERVENTIONS:
Device: rTMS on ipsilesional M1
Device: tDCS on contralesional M1
  Arms: Dual-mode stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) or transcranial direct current stimulation (tDCS) has been used for the modulation of stroke patients' motor function by altering the cortical excitability. Recently, more challenging approaches, such as stimulation of two or more sites or use of dual modality have been studied in stroke patients. In this study, simultaneous stimulation using both rTMS and tDCS (dual-mode stimulation) over bilateral primary motor cortices (M1s) was investigated to compare its modulatory effects with single rTMS stimulation in subacute stroke patients.

DETAILED DESCRIPTION:
Investigators assessed each patient's motor function using the Fugl-Meyer Assessment (FMA) score and acquired their resting-state fMRI (rs-fMRI) data at two times: prior to stimulation and 2 months after stimulation. Changes in rs-fMRI network measures were investigated between groups.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke patients
* Subacute stage (less than 4 weeks)
* Total Fugl-Meyer Assessment (FMA) score under 84

Exclusion Criteria:

* Major active neurological disease or psychiatric disease
* A history of seizure
* Metallic implants in their brain

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Neuroimaging Assessment | Change from baseline resting-state brain network at 8 weeks after intervention
  Resting-state fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Park E, Lee A, Chang WH, Kim DS, Shin YI, Kim YH. Modulating Brain Connectivity by Simultaneous Dual-Mode Stimulation over Bilateral Primary Motor Cortices in Subacute Stroke Patients. Neural Plast. 2018 Feb 13;2018:1458061. doi: 10.1155/2018/1458061. eCollection 2018. PMID 29666636

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03279640/Prot_SAP_000.pdf